CLINICAL TRIAL: NCT02270489
Title: A Randomized, Placebo-controlled, Parallel Group, Patient-blind, Phase I Study Assessing the Safety and Exploring the Immunogenicity/Therapeutic Activity of AFFITOPE® PD01A and PD03A in Patients With Early Multiple System Atrophy
Brief Title: Study Assessing Safety and Therapeutic Activity of AFFITOPE® PD01A and PD03A in Patients With Early MSA
Acronym: AFF009
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affiris AG (Industry)
Collaborators: University Hospital, Bordeaux (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Forschungszentrum Juelich (Other); University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFFiRiS 009; 2014-000567-40 (EudraCT Number)
Record Dates: First submitted 2014-09-04; First posted 2014-10-21 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Multiple System Atrophy; Neurodegenerative Diseases
MeSH Terms: conditions — Multiple System Atrophy; Neurodegenerative Diseases | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AFFITOPE® PD01A + Adjuvant (Experimental): 4 injections of 75µg AFFITOPE® PD01A/ adjuvanted, once every 4 weeks
  1 boost immunization 36 weeks after first injection
  Interventions: Biological: AFFITOPE® PD01A + Adjuvant
- AFFITOPE® PD03A + Adjuvant (Experimental): 4 injections of 75µg AFFITOPE® PD03A/ adjuvanted, once every 4 weeks
  1 boost immunization 36 weeks after first injection
  Interventions: Biological: AFFITOPE® PD03A + Adjuvant
- Adjuvant without active component (Placebo Comparator): 4 injections of Placebo once every 4 weeks
  1 administration 36 weeks after first injection
  Interventions: Biological: Adjuvant without active component

INTERVENTIONS:
Biological: AFFITOPE® PD01A + Adjuvant — s.c. injection
  Arms: AFFITOPE® PD01A + Adjuvant
Biological: AFFITOPE® PD03A + Adjuvant — s.c. injection
  Arms: AFFITOPE® PD03A + Adjuvant
Biological: Adjuvant without active component — s.c. injection
  Arms: Adjuvant without active component

SUMMARY:
This is a randomized controlled parallel Group phase I study to investigate the safety and immunological/ therapeutic activity of two new vaccines, AFFITOPE® PD01A and AFFITOPE® PD03A, given to patients with early Multiple System Atrophy (MSA).

In total 30 patients are planned to be enrolled in the study: 12 patients in each treatment arm who will receive either 75µg AFFITOPE® PD01A (with adjuvant) or 75µg AFFITOPE® PD03A (with adjuvant) and 6 patients in the control group who will receive the reference substance (Placebo). Over a study duration of 52 weeks, the study participants will receive 4 injections as basic immunization in a 4-weekly interval and 1 boost immunization 36 weeks after the first injection. Male and female patients aged 30 to 75 years can participate in the trial. 2 study sites in France (Bordeaux and Toulouse) will be involved.

AFF009 is part of the project SYMPATH funded by the European Commission (FP7-HEALTH-2013-INNOVATION-1 project; N° HEALTH-F4-2013-602999).

ELIGIBILITY:
Inclusion Criteria:

* Possible or probably MSA diagnosis (MSA-P or MSA-C) according to Gilman 2008 consensus criteria
* Onset of MSA symptoms less than 4 years
* Participants with an anticipated survival of at least 3 years in the opinion of the PI
* Written informed consent obtained prior to study entry
* MSA patient > 30 and < 75 years of age at time of study entry
* Female patients of childbearing potential using a medically accepted contraceptive method
* Stable medication for MSA symptoms (Levodopa, Dopamine agonists, Midodrine, Fludrocortisone, monoamine oxidase-B and Catechol-O-methyltransferase inhibitors; Antidepressants, Laxatives, NSAIDs or paracetamol as basic medication for pain in the musculoskeletal system)

Exclusion Criteria:

* Pregnant or lactating women
* Sexually active women of childbearing potential not using a medically accepted birth control method
* Patients with dementia (MOCA at Screening < 21)
* Speech impairment as assessed by a score of ≥ 3 on UMSARS question 1
* Swallowing impairment as assessed by a score of ≥ 3 on UMSARS question 2
* Impairment in ambulation as assessed by a score of ≥ 3 on UMSARS question 7
* History or evidence of any other central nervous system disorder like stroke, angioma and other relevant neurological diseases
* History of malignancy other than skin cancer during the last 5 years (if considered to be cured, patient might be included)
* Active or passive vaccination 4 weeks before the first vaccination on Day 0 and during the main study period ending on Day 280. Emergency vaccinations are acceptable
* Use of any other investigational or non-registered drug or vaccine in addition to the study vaccine during the entire study period
* Subjects participating or have participated in another interventional clinical trial within 60 days prior to baseline
* Blood donation within 4 weeks prior to first vaccination.
* History of autoimmune diseases, severe hypersensitivity reactions and anaphylaxis, allergic bronchial asthma and severe allergic rhinoconjunctivitis
* Known hypersensitivity or allergic reaction to one of the components of the vaccine
* A family history of congenital or hereditary immunodeficiency
* Administration of chronic (defined as more than 14 days) immunosuppressant or other immune-modifying drugs within six months before first vaccination and during the entire study period. For corticosteroids like prednisone or equivalent ≥ 0.05 mg/kg/day. Topical and inhaled steroids are allowed
* Intake of non steroidal anti-inflammatory drugs (NSAIDs) or paracetamol more than the basic medication for pain in the musculoskeletal system within three days prior to a vaccination with AFFITOPE® PD01A or AFFITOPE® PD03A or Placebo
* If a patient shows an acute febrile infection (≥ 37.8° Celsius) on the day of vaccination, administration of Investigational Medicinal Product (IMP) should be postponed until resolution of the infection
* Infection with the human immunodeficiency virus (HIV, a negative test result within 30 days before screening is acceptable), Hepatitis B (HBsAg) or Hepatitis C
* Significant systemic illness (e.g. chronic renal failure, chronic liver disease, poorly controlled diabetes, poorly controlled congestive heart failure and/or other deficiencies), if considered relevant by the investigator
* Venous status rendering it impossible to place an i.v. access
* Contraindications for MRI and lumbar puncture
* Not able to understand and comply with protocol requirements, instructions, protocol-stated restrictions
* Unwilling to provide informed consent. Exceptions for patients who are physically not able to provide written informed consent (e.g. legal representative, consent via voce with witness)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
Number of patients who withdraw due to Adverse Events (AEs) | 12 months
Occurrence of Adverse Events and Serious Adverse Events | 12 months
  Evaluation of Adverse Events and Serious Adverse Events in regards to autoimmune reactions
Physical Examination | 12 months
  New findings or change in pre-existing findings assessed in physical examinations over time (study period)
Vital signs | 12 months
  Change in vital signs. The Evaluation includes the changes in blood pressure, heart rate, respiratory rate and Body temperature over time (measured at each visit).
Safety related evaluation of MRI results of patients' brain after visit 5 and visit 8 compared to baseline | 12 months
  Safety measures will e.g. include the occurrence of inflammatory reactions (meningoencephalitis), new/changed hemorrhages and lacunar infarcts.
Clinical significance/ changes in laboratory parameters over time (study period) | 12 months
  Laboratory assessment includes hematology, biochemistry, coagulation, serology and urinanalysis
Body mass | 12 months
  Change of Body mass over time (study period)
Neurological Examination | 12 months
  New findings or change in pre-existing findings assessed in neurological examinations over time (study period)

SECONDARY OUTCOMES:
Immunological activity of AFFITOPE® vaccines PD01A and PD03A. | 12 months
  Titer of vaccination induced antibodies directed towards vaccine components, alpha- and beta synuclein
Change in motor symptoms at Visit 5 and Visit 8 compared to baseline | 12 months
  Change in Motor symptoms: UMSARS II (Unified Multiple System Atrophy Rating Scale), CGI (Clinical Global Impression Improvement scale)
Change in non-motor symptoms at Visit 5 and Visit 8 compared to baseline | 12 months
  Change in non-motor symptoms: UMSARS I and IV, GDS (Geriatric Depression Scale), COMPASS 31 (Composite Autonomic Symptom Score), MSA-QoL (MSA- Quality of life scale), MOCA (Montreal cognitive assessment), autonomic testing of cardiovascular function

CONTACTS AND LOCATIONS:
Overall Officials: Wassilios Meissner, MD, PhD, Principal Investigator — University Hospital Bordeaux (Pellegrin Hospital), Bordeaux 33076, France
Locations (2):
- France (2):
  - University Hospital Bordeaux (Pellegrin Hospital), Bordeaux
  - University Hospital Toulouse, Toulouse

REFERENCES:
- [Derived] Meissner WG, Traon AP, Foubert-Samier A, Galabova G, Galitzky M, Kutzelnigg A, Laurens B, Luhrs P, Medori R, Peran P, Sabatini U, Vergnet S, Volc D, Poewe W, Schneeberger A, Staffler G, Rascol O; AFF009 Study Investigators. A Phase 1 Randomized Trial of Specific Active alpha-Synuclein Immunotherapies PD01A and PD03A in Multiple System Atrophy. Mov Disord. 2020 Nov;35(11):1957-1965. doi: 10.1002/mds.28218. Epub 2020 Sep 3. PMID 32882100